CLINICAL TRIAL: NCT02580695
Title: A Phase I/II, Randomized, Double-blind, Controlled Study to Assess Safety and Efficacy of Umbilical Cord-derived Mesenchymal Stromal Cells (UC-MSCs) in Patients With Knee Osteoarthritis
Brief Title: A Study to Assess Safety and Efficacy of Umbilical Cord-derived Mesenchymal Stromal Cells in Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Francisco Espinoza, MD (Other)
Responsible Party: Sponsor-Investigator, Francisco Espinoza, MD, Alternative Investigator, Universidad de los Andes, Chile
Organization: Universidad de los Andes, Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C4COA01
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical-cord mesenchymal stromal cells (Experimental): Umbilical-cord mesenchymal stromal cells (UC-MSCs)
  Allogeneic UC-MSCs 20 x 10e6 diluted on 3 mL of saline solution + 5% of Plasma AB
  Arm 2a: single infusion group. UC-MSCs at 0 month
  Arm 2b: double infusion group. UC-MSCs at 0 and 6 months
  Interventions: Biological: umbilical-cord mesenchymal stromal cells
- Hyaluronic Acid (HA) (Active Comparator): Drug: Hyaluronic Acid 3 mL of HA intra-articular injection at baseline and 6 months
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: umbilical-cord mesenchymal stromal cells — Intra-articular knee injection of UC-MSC 20x10e6 at 0 and 6 months
  Other Names: UC-MSCs
  Arms: Umbilical-cord mesenchymal stromal cells
Drug: Hyaluronic Acid — Intra-articular knee injection of Hyaluronic Acid (3ml) at 0 and 6 months
  Other Names: Durolane
  Arms: Hyaluronic Acid (HA)

SUMMARY:
Knee-osteoarthritis (OA) is a common and disabling problem, that represents a global health issue since none of the current therapies are truly disease modifying. The use of mesenchymal stem cells (MSCs) in OA-preclinical models has been associated with a reduction in cartilage degradation, the attenuation of bone sclerosis and an effective anti-inflammatory response. Investigators have designed a randomized phase I/II placebo controlled trial of UC-MSCs in knee OA. Outcomes will be evaluated at 12 months, comparing monodosis versus double intra-articular injection, re-randomized at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Knee OA, Kellgren and Lawrence grade I, II, III on plain Rx films.
* Chondromalacia patella grade I-III on knee MRI. With or without meniscal tear.
* Stable knee and normal clinical exam of involved extremity
* Written informed consent for patients.

Exclusion Criteria:

* Bilateral symptomatic knee OA
* Local or systemic infection.
* Active neoplasia or immunosuppressive state
* Pregnancy or Breastfeeding
* Body Mass Index ≥ 30
* Presence of Pacemaker or Lower extremity metal implant
* Anticoagulant treatment other than aspirin.
* Recent use of oral (previous month) or intra-articular (previous 3 months) corticosteroids
* Concomitant inflammatory joint disease (cristal, connective tissue disease)
* Valgus (>10o) or Varus (>5o) deformity of involved extremity
* Condilar or Tibial plateau Generalized Bone Marrow edema on MRI
* Significant symptomatic hip or spine disease
* Significant abnormality in baseline lab tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience an adverse event | 12 months
  according to National Cancer Institute Common Terminology Criteria for Adverse Effects (NCI-CTCAE)

SECONDARY OUTCOMES:
Physical function improvement measured by WOMAC OA index | 12 months
Change in pain density measured by Visual analogue scale (VAS) | 12 months
QoL improvement measured by SF-36 | 12 months
Changes in WORMS scale measured by knee MRI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Matas, MD, Principal Investigator — Universidad de Los Andes
Locations (1):
- Clinica Universidad de los Andes, Santiago, Chile